CLINICAL TRIAL: NCT03070015
Title: The Effects of a Commercially Available Weight Loss Program on Body Weight in Overweight Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrisystem, Inc. (Industry)
Collaborators: The Center for Applied Health Sciences (Unknown); Omega Statistics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTR001-2015
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Overweight and Obesity; Weight Loss
Keywords: Weight Loss; Obesity; Overweight
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrisystem (Experimental): All subjects received Nutrisystem pre-packaged, portion-controlled foods and followed the Nutrisystem program for a total of 12 weeks (4 weeks for Part A, and an additional 8 weeks for Part B)
  Interventions: Behavioral: Nutrisystem
- Self-Directed DASH (Active Comparator): All subjects provided publically available information on the DASH diet and a sample meal plan. Subjects were instructed to follow a reduced calorie DASH diet meal plan on their own for 4 weeks (Part A only).
  Interventions: Behavioral: Self-Directed DASH

INTERVENTIONS:
Behavioral: Nutrisystem — The Nutrisystem Diet was 1000 kcal/day for week 1,and 1200 calories/day for women and 1500 calories/day for men after week 1.Subjects with BMI > 40 added 200 extra calories/day through grocery food add-ins.Subjects received 7 breakfast,7 lunches,7 dinners, and 14 shakes for week 1.Subjects added in vegetables & no-calorie beverages in week 1.After week 1,Nutrisystem provided 7 breakfasts,6 lunches,6 dinners, and 7 (women) or 14 (men) snacks/week.Subjects prepared 1 lunch & 1 dinner on their own weekly. Guidelines were given to allow subjects to select foods that fit within plan guidelines (~50% kcal from carbohydrate,~25% from protein,~25% from fat). Nutrisystem foods were about 60% of kcal target; grocery additions made the balance.Subjects received guidance as typical on Nutrisystem throughout the study period.Subjects were encouraged to call Nutrisystem counselors. Subjects randomized to this participated in Part A (4 weeks) and Part B (additional 8 weeks) of the study.
  Arms: Nutrisystem
Behavioral: Self-Directed DASH — The self-directed Dietary Approaches to Stop Hypertension group received instruction/education with handouts & sample meal plans, which met guidelines for DASH. All subjects followed a 1000 kcal/day DASH diet for week 1. After week 1, women ate 1200 kcal/day & men ate 1500 kcal/day. Subjects with BMI >40 added an extra 200 kcal/day. Subjects randomized to this group received one additional educational session beyond the Randomization visit on how to follow their prescribed meal plan. Subjects in this group only participated in Part A (4-weeks) of the study.
  Arms: Self-Directed DASH

SUMMARY:
The primary purpose of this study (Part A) is to assess changes in body weight and body circumference parameters that are achievable after 4 weeks on the Nutrisystem program compared to a self-directed diet (i.e. Dietary Approaches to Stop Hypertension or DASH). In Part B, subjects on the Nutrisystem program will be given the option to continue the program for another 8 weeks.

DETAILED DESCRIPTION:
A randomized, controlled, parallel study design with two parts (Part A and Part B). Study visits include Screening, Randomization, and Weeks 1, 2, 3 and 4. Week 4 serves also as the closeout study visit for Part A. Subjects randomized to the intervention group (i.e., Nutrisystem group) will continue the program for an additional 8 weeks, and include additional study visits at week 8 and 12.

Eighty-four (N=84) healthy men and women, matched paired for BMI, will be randomized into one of two groups for 28 days (4 weeks): Nutrisystem program or a self-directed Dietary Approaches to Stop Hypertension ("DASH"). All subjects in the Nutrisystem group who complete Part A will continue on the Nutrisystem program for an additional 8 weeks (Part B).

Daily energy intake targets for each group will include a 1000 kcal/day diet for both women and men during the first week. After the first week women will follow a 1200 kcal/day diet and men will follow a 1500 kcal/day diet. Subjects with BMI > 40 will add approximately 200 additional calories to their diet each day.

Body weight and body circumference (Waist, Hip, Chest, Arm & Thigh and Sum of the 5) measures were obtained at baseline and weeks 1, 2, 3, 4 (Part A). And at weeks 8 and 12 for the Nutrisystem group (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 19-70 years of age, inclusive.
* Subject has a BMI of 25.00 to 44.99 kg/m2 at the Screening visit.
* Subject is a non-smoker.
* Female study participants ages 19-49 must be on a steady dose of oral contraceptives (OCA) [to reduce weight variability secondary to changes that occur with the luteal phase of menses]. Stable dose was defined as same dose for at least past 90 days. Female study participants that are 50 or over who are not currently on birth control but are weight stable for at least the prior three months were enrolled.
* Subject is willing to follow study program instructions, including avoidance of all non-study-related food and beverages.
* Subject is willing and able to comply with the visit schedule.
* Subject agrees to follow the instructions and meal plans per the randomization into Nutrisystem or Self-Directed.
* Subject agrees to follow the physical activity recommendations as outlined in each plan.
* If a premenopausal female, subject has a history of regular menstrual cycles that range in length from 21 to 35 d, where applicable.
* Judged to be in good health on the basis of medical history and screening laboratory assessments.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

* Females with prior diagnosis of premenstrual syndrome or Premenstrual dysphoric disorder (PMDD).
* Subject has an abnormal laboratory test result of clinical significance at the Screening visit that upon re-testing has not normalized (per physician discretion).
* Subject has had a weight loss or gain ≥10 lb (4.5 kg) in the three (3) months prior to Visit 1 (Week -1).
* Subject has used weight loss medications within the past three months of Screening visit.
* Subject has dietary tendencies that may be representative of disordered eating (in the opinion of the Investigator).
* Subject has a known allergy, sensitivity, or intolerance to the study foods or any ingredients of the study menu provided.
* Subject has previously been diagnosed diabetes mellitus (type 1 or type 2) or fasting glucose ≥126 mg/dL at the screening visit.
* Subject is on thyroid medication at a dose that is not considered stable. Stable is same dose consistently for at least 90 days.
* Subject has used any prescription weight loss medications within three months prior to Screening Visit, and any dietary supplements or programs intended to alter body weight within the last four weeks.
* Subject uses hypoglycemic medications (with or without diagnosis of diabetes, e.g. metformin for PCOS is exclusionary) or dietary supplements that may affect carbohydrate metabolism.
* Subject has used any prescription Corticosteroids (oral or systemic) within past three months.
* Subjects using medications and dietary supplements likely to markedly affect appetite or metabolic rate (e.g., beta-blockers) may be excluded, based on the judgment of the Investigator (with washout prior to study randomization).
* Subject has a history or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurologic disorders.
* Subject has an active gastrointestinal disorder such as peptic ulcer disease or malabsorption syndrome (mild lactose intolerance or gastroesophageal reflux diseases are acceptable).
* Subject has an active infection or sign/symptoms of an infection. The randomization visit will be re-scheduled to allow subject to be symptom-free of any type of systemic infection for at least 5 days.
* Subject has a history of gastrointestinal surgery that is known to affect nutrient absorption or body weight.
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at the Screening visit.
* Subject has a history or presence of cancer in the prior 5 years, except for non-melanoma skin cancer.
* Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception (double-barrier method) throughout the study period. The method of contraception must be recorded in the source document.
* Subject is a premenopausal female using a form of hormonal contraception that does not result in a normal menstrual cycle, including a regular menses period.
* Subject has a recent history of (within 12 months of Visit 1, Week -1) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Subject has been hospitalized within the past one-year for any mental or emotional illness.
* Exposure to any non-registered drug product within 30 d prior to the screening visit.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Body Weight | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in body weight from baseline (week 0) to each post-randomization visit (week 1, 2, 3, and 4 for Parts A & B; plus week 8, 12 for Part B)

SECONDARY OUTCOMES:
Waist Circumference | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in waist circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4 for Parts A & B; plus week 8, 12 for Part B)
Hip Circumference | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in hip circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4 for Parts A & B; plus week 8, 12 for Part B)
Chest Circumference | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in chest circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4 for Parts A & B; plus week 8, 12 for Part B)
Arm Circumference | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in arm circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4 for Parts A & B; plus week 8, 12 for Part B)
Thigh Circumference | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in thigh circumference from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4 for Parts A & B; plus week 8, 12 for Part B)
Sum of the 5 Body Circumferences | up to 4 weeks (Part A); up to 12 weeks (Part B)
  Change in Sum of 5 body circumferences (waist, hip, chest, arm, thigh) from baseline (week 0) to each post-randomization visit (week 1, 2, 3, 4 for Parts A & B; plus week 8, 12 for Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Tim N Ziegenfuss, Ph.D., FISSN, CSCS, Principal Investigator — The Center for Applied Health Sciences

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.